CLINICAL TRIAL: NCT01558219
Title: Open, Single-arm, Multicenter, Phase II Trial Investigating the Safety of Biweekly Cabazitaxel in Metastatic Castration Resistant Prostate Cancer Patients Previously Treated With a Docetaxel-containing Regimen
Brief Title: Second-line Chemotherapy in Castration Resistant Prostate Cancer
Acronym: ProstyII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Helsinki University Central Hospital (Other); Turku University Hospital (Other Government); Kuopio University Hospital (Other); Seinajoki Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-003156-39
Record Dates: First submitted 2011-11-25; First posted 2012-03-20 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Metastatic Prostate Cancer
Keywords: Metastatic prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- acitive anticancer drug (Experimental): single cytostatic agent, cabazitaxel every second week in the treatment of castration resistant metastatic prostate cancer after docetaxel
  Interventions: Drug: cabacitaxel

INTERVENTIONS:
Drug: cabacitaxel — Jevtana® (cabazitaxel) 16 mg/m2 IV in 1 hour on day 1 given every second week

SUMMARY:
This study is designed to evaluate the safety of biweekly cabazitaxel for the treatment of metastatic castration resistant prostate cancer (mCRPC) patients previously treated with docetaxel containing regimen. The primary endpoint is safety. Secondary endpoints include time to treatment failure, response rate, overall survival and quality of life.

DETAILED DESCRIPTION:
The objective of this study is to explore new, biweekly schedule of cabazitaxel in metastatic castration resistant prostate cancer patients. A previous study has shown that the biweekly administration of docetaxel in 1st line setting of mCRPC is better tolerated than docetaxel administered every three weeks. Also, the efficacy of biweekly docetaxel was better than three-weekly docetaxel and biweekly dosing presented a significant overall survival benefit (ASCO 2011, Kellokumpu-Lehtinen et al. As the occurrence of neutropenia in the TROPIC trial was rather high, the hypothesis is to reduce the incidence of severe adverse events by administrating cabazitaxel more frequently, yet maintaining the same dose intensity as in every three weeks´ dosing schedule.

This study is designed to evaluate the safety of biweekly cabazitaxel for the treatment of 60 patients with metastatic castration resistant prostate cancer (mCRPC) patients previously treated with docetaxel containing regimen.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic castration resistant prostate cancer
* Disease progression during or after docetaxel-containing regimen for mCRPC
* Surgical or medical castration
* WHO performance status < 2
* Age > 18 years
* Adequate bone marrow, liver and renal functions:

Hematology:

* neutrophils > 1.5 x 109/ l
* hemoglobin > 100 g/l
* platelets > 100 x 109/l

Hepatic and renal functions:

* total bilirubin <1 x ULN
* ALAT and ASAT < 2.5 x ULN, alkaline phosphate <6 x ULN.In the presence of extensive bone disease, alkaline phosphate > 6 x ULN is accepted
* creatinine < 1.5 x ULN (ie NCI CTC-AE grade < 1)

Exclusion Criteria:

* Prior surgery, radiation, chemotherapy, or other anti-cancer therapy within 4 weeks prior to enrollment
* Prior therapy with radioisotopes
* Other malignant disease (except superficial non-melanoma skin cancer) within the past 5 years
* Serious liver disease
* History of severe hypersensitivity reaction (grade > 3) to polysorbate 80 containing drugs
* Concurrent or planned treatment with potent inhibitors or inducers of cytochrome P450 3A4/5 (a one week wash-out period is necessary for patients who already are on these treatments)
* Other serious illness or medical condition:
* Serious cardiac disease; ischemic or thromboembolic cardiac disease, pulmonary emboli, cardiac infarction within 12 months
* Active infection
* Active peptic ulcer, uncontrolled diabetes mellitus or other contraindications for the use of corticosteroids
* Auto-immune disease (lupus, scleroderma, rheumatoid polyarthritis)
* Active grade > 2 polyneuropathy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerabilty | every 2 weeks
  NCI CTC-AE version 4 Adverse events in every organ systems and laborotory values (Grades from 0 to 5, 0=no adverse events, 5= dead)from baseline up to the end of the treatment

SECONDARY OUTCOMES:
Response rate | PSA every 6 week, tumor assesment every 12 week
  Recist version 1.1 (response evaluation of solid solid tumors; Eisenhauer et al. JCO 2009;45:228-247)

CONTACTS AND LOCATIONS:
Overall Officials: Pirkko-Liisa I kellokumpu-Lehtinen, MD, PhD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland